CLINICAL TRIAL: NCT00940797
Title: Effect of DMMET-01 on Insulin Sensitivity in Naive Type 2 Diabetes Patients by Glucose CLAMP Technique
Brief Title: Effect of DMMET-01 on Insulin Sensitivity in Naive Type 2 Diabetes Patients (CLAMP)
Acronym: DMMETclamp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Jorge González Canudas/Medical director, Silanes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-1099/2008; SIL-DMMETClamp
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Type 2
Keywords: diabetes; Type 2; monotherapy; antidiabetics; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMMET-01 (Experimental)
  Interventions: Drug: DMMET-01
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMMET-01 — 60 days: 30 days; dose 1050.6 mg per day (before dinner)+ 30 days; dose 1050.6 mg twice a day 30 more days (before breakfast ando before dinner)
  Arms: DMMET-01
Drug: Placebo — 60 days: 30 days placebo once a day (before dinner) + 30 days twice a day (before breakfast and before dinner)
  Arms: Control

SUMMARY:
The aim of this study is to determine the effect of DMMET-01 on insulin sensitivity by Glucose CLAMP technique in Mexican type 2 diabetes patients, after 2 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 40 to 60 years
* With type 2 diabetes evolution < 5 years without pharmacological treatment 1 month prior to the screening
* Fasting glucose = 130-200 mg/dL
* AIc of 7% to 9%
* Blood pressure < 140/80 mmHg
* Ability to communicate and meet the requirements of the study
* Signed Written Informed Consent before to conducting any study
* Body mass index (BMI) of 25 kg/m2 to 35 Kg/m2

Exclusion Criteria:

* Suspected or confirmed pregnancy
* Nursing
* Inability to secure the non-pregnant during the study duration
* Hypersensitivity to any biguanides
* Use of an investigational drug within 30 days prior to the screening
* Liver failure, heart failure, kidney failure or thyroid disease
* Periods of acute or chronic diarrhea or vomiting
* Chronic hepatic disease
* Total Cholesterol > 300 mg/dL
* Triglycerides > 400 mg/dL

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 months

SECONDARY OUTCOMES:
Insulin, fasting glucose, HbA1c | 2 months
Adverse Events | 3 months
Creatinine, Total Cholesterol, HDL, Triglycerides, Uric acid, AST, ALT, FA, DHL | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A González, MD, Study Director — Laboratorios Silanes S.A. de C.V.; Manuel Gonzalez, PHD, Study Chair — University of Guadalajara; Esperanza Martínez, PHD, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, México, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Aguilar-Salinas CA, Velazquez Monroy O, Gomez-Perez FJ, Gonzalez Chavez A, Esqueda AL, Molina Cuevas V, Rull-Rodrigo JA, Tapia Conyer R; Encuesta Nacional de Salud 2000 Group. Characteristics of patients with type 2 diabetes in Mexico: Results from a large population-based nationwide survey. Diabetes Care. 2003 Jul;26(7):2021-6. doi: 10.2337/diacare.26.7.2021. PMID 12832306
- [Background] González-Ortiz M, Martínez-Abundis E. Síndrome de resistencia a la insulina. En, Diabetes mellitus. Islas-Andrade S, Revilla-Monsalve C. McGrawHill-Interamericana. 3a. edición. México, 2005. ISBN p. 203-14.
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Derived] Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Ramos-Zavala MG, Barrera-Duran C, Gonzalez-Canudas J. Effect of metformin glycinate on glycated hemoglobin A1C concentration and insulin sensitivity in drug-naive adult patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2012 Dec;14(12):1140-4. doi: 10.1089/dia.2012.0097. Epub 2012 Sep 13. PMID 22974412